CLINICAL TRIAL: NCT02202187
Title: A Randomized, Single Blind, Placebo Controlled Study to Evaluate Safety, Tolerability, and Pharmacokinetics of Single Escalating Oral Doses of GSK2140944 in Healthy Adult Subjects
Brief Title: A Single Oral Escalating Dose Study of GSK2140944 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 114595
Record Dates: First submitted 2012-03-29; First posted 2014-07-28 (Estimated); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: Infections, Respiratory Tract
MeSH Terms: conditions — Respiratory Tract Infections | interventions — gepotidacin

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- GSK2140944 (Experimental): Dose range 100mg to 3000mg single dose
  Interventions: Drug: GSK2140944
- Matching Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: GSK2140944 — Investigational Study Drug
  Arms: GSK2140944
Other: Placebo — Placebo
  Arms: Matching Placebo

SUMMARY:
GSK2140944 belongs to the Bacterial Type II Topoisomerase Inhibitor (BTI) class of antibiotics. GSK2140944 has demonstrated in vitro and in vivo activity against Gram positive including methicillin resistant Staphylococcus aureus (MRSA) and Gram-negative pathogens associated with respiratory tract, skin and soft tissue infections including isolates resistant to existing classes of antimicrobials. This is a First Time in Human (FTIH) study to assess the safety, tolerability, and pharmacokinetics of single oral doses of GSK2140944 in healthy volunteers. This study will be a single-blind, randomized, placebo-controlled, dose-rising study in healthy subjects. The proposed single doses will range from 100 mg to 3000 mg.

DETAILED DESCRIPTION:
GSK2140944 belongs to the Bacterial Type II Topoisomerase Inhibitor (BTI) class of antibiotics which is being developed for treatment of Gram positive [including methicillin resistant Staphylococcus aureus (MRSA)] and Gram-negative pathogens associated with respiratory tract and skin and soft tissue infections including isolates resistant to existing classes of antimicrobials.

Study BTZ114595 will be the first administration of GSK2140944 in humans. This study will examine the safety, tolerability, and pharmacokinetics of escalating single oral doses of GSK2140944. The predicted clinical target for efficacy, based on preclinical efficacy models, is an AUC(0-24) of 16-30 μg.h/mL. This study aims to explore the safety and tolerability at and above target exposures in order to establish a therapeutic window for this compound.

This study will investigate the safety, tolerability, and pharmacokinetics of escalating single oral doses of GSK2140944.

This will be a randomized, placebo-controlled, single-blind study to determine safety, tolerability, and single dose pharmacokinetic (PK) profile of GSK2140944 in healthy subjects.

The projected single escalating doses of GSK2140944 will range from a starting dose of 100 mg to a maximum dose of 3000 mg. The current plan is to administer the study drug after an overnight fast, but based on emerging PK and safety data, it may be necessary to administer the study drug under fed state to better understand safety, tolerability or PK of GSK2140944. Any decision to remove or modify fasting requirements will be made by the GSK Study Team and the investigator based on joint review of the emerging safety, tolerability and preliminary pharmacokinetic data from prior dose-levels.

ELIGIBILITY:
Inclusion Criteria:

* AST, ALT, alkaline phosphatase and bilirubin ≤ 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%)
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Male or female ranging from 18 to 60 years of age, at the time of signing the informed consent. Female subject must be of non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and estradiol < 40 pg/mL (<147 pmol/L) is confirmatory]. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods in Section 8.1 if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least 2-4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method.
* Body weight ≥ 50 kg and BMI within the range 19 - 31 kg/m2, inclusive.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* QTcF < 450 msec, or QTc < 480 msec in subjects with Bundle Branch Block., at screening.

Exclusion Criteria:

* Any clinically significant central nervous system (e.g., seizures), cardiac, pulmonary, metabolic, renal, hepatic or gastrointestinal conditions or history of such conditions that, in the opinion of the investigator may place the subject at an unacceptable risk as a participant in this trial or may interfere with the absorption, distribution, metabolism or excretion of drugs.
* A positive urine test for drugs of abuse or alcohol (or alcohol breath test) at screening.
* A screening urinalysis positive for protein or glucose (greater than "trace" findings of protein or glucose).
* Positive for Human Immunodeficiency Virus (HIV) antibody, hepatitis B virus surface antigen, or hepatitis C virus antibody at screening.
* History of drug abuse within 6 months of the study.
* History of smoking or use of nicotine containing products within 3 months of screening, or a positive urine cotinine indicative of smoking at screening.
* History of regular alcohol consumption exceeding an average weekly intake of greater than or equal to 21 units for men/14 units for women or an average daily intake of greater than or equal to 3 units for men/2 units for women. One unit is equivalent to a 285 mL glass of full strength beer or 425 mL schooner of light beer or 1 (30 mL) measure of spirits or 1 glass (100 mL) of wine.
* The subject has participated in a clinical trial and has received a drug or a new chemical entity within 30 days or 5 half-lives, or twice the duration of the biological effect of any drug (whichever is longer) prior to the first dose of current study medication.
* Use of prescription or non-prescription drugs, including vitamins above the recommended daily intake (National Health and Medical Research Council in Australia guideline), herbal and dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study medication, or use of St. John's Wort within 14 days prior to the first dose of study medication. By exception, the volunteer may take paracetamol or acetaminophen (≤ 2 grams/day) or ibuprofen (1600 mg/day) up to 48 hours prior to the first dose of study medication. However, the investigator and study team can review medication use on a case by case basis to determine if its use would compromise subject safety or interfere with study procedures or data interpretation.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice, pummelos, exotic citrus fruits or grapefruit hybrids or fruit juices containing such products for 7 days prior to administration of study medication.
* Donation of blood in excess of 550 mL within 12 weeks prior to dosing.
* An unwillingness of male subjects to abstain from sexual intercourse with pregnant or lactating women, or an unwillingness of male subjects to use a condom and spermicide, in addition to having their female partner use another form of contraception such as an IUD, diaphragm with spermicide, oral contraceptives, injectable progesterone, subdermal implants or a tubal ligation, if engaging in sexual intercourse with a female partner who could become pregnant. This criterion must be followed from the time of study medication administration and until 84 days after study medication administration.
* History of sensitivity to any of the study medications or components thereof or a history of drug or other allergy that, in the opinion of the physician responsible, contraindicates their participation.
* History of sensitivity to heparin or heparin-induced thrombocytopenia (if the clinical research unit uses heparin to maintain intravenous cannula patency).
* An unwillingness to comply with lifestyle and/or dietary restrictions as described in Section 8.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2011-09-26 (Actual); Primary Completion 2012-02-15 (Actual); Study Completion 2012-02-15 (Actual)

PRIMARY OUTCOMES:
GSK2140944 clinical safety data assessed as change from baseline in 12-lead ECG | Day 1, Day 2, Day 3 and at the Follow-up visit
  12-lead ECGs will be obtained at each timepoint using an ECG machine, after the subject has rested in the supine position for at least 10 minutes
GSK2140944 clinical safety data from dual-lead cardiac monitoring | Day -1, Day 1
  Continuous dual-lead cardiac monitoring will be obtained at each timepoints using an ECG machine
GSK2140944 clinical safety data assessed as change from baseline in clinical laboratory tests | Day -1, Day 2, Day 3 and the Follow-up visit
  Clinical laboratory assessments will include hematology, clinical chemistry, routine urinalysis and additional parameters
GSK2140944 clinical safety data assessed as by number of adverse events (AE) | Up to the Follow-up visit
  Safety and tolerability parameters will include recording of AEs, throughout the study
GSK2140944 clinical safety data assessed as change from baseline in blood pressure | Day -1, Day 1, Day 2, Day 3 and the Follow-up visit
  Vital sign measurements will include systolic and diastolic blood pressure
GSK2140944 clinical safety data assessed as change from baseline in heart rate | Day -1, Day 1, Day 2, Day 3 and the Follow-up visit
  Vital sign measurements will include pulse rate

SECONDARY OUTCOMES:
Pharmacokinetic parameter: AUC(0-t) following single dose of GSK2140944 | Up to Day 4
  Pharmacokinetic data will include area under the concentration-time curve from time zero (pre-dose) to last time of quantifiable concentration (AUC(0-t)) following single dose of GSK2140944
Pharmacokinetic parameter: AUC(0-infinity) following single dose of GSK2140944 | Up to Day 4
  Pharmacokinetic data will include area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time (AUC(0-infinity)) following single dose of GSK2140944
Pharmacokinetic parameter: Cmax following single dose of GSK2140944 | Up to Day 4
  Pharmacokinetic data will include maximum observed concentration (Cmax) following single dose of GSK2140944
Pharmacokinetic parameter: tmax following single dose of GSK2140944 | Up to Day 4
  Pharmacokinetic data will include time of occurrence of Cmax (tmax) following single dose of GSK2140944
Pharmacokinetic parameter: t1/2 following single dose of GSK2140944 | Up to Day 4
  Pharmacokinetic data will include terminal phase half-life (t1/2) following single dose of GSK2140944
To assess preliminary dose proportionality using PK parameter AUC(0-infinity) following single dose of GSK2140944 | Up to Day 4
  Preliminary dose proportionality will be assessed using PK parameter (AUC(0-infinity)) following single dose of GSK2140944
To assess preliminary dose proportionality using PK parameter Cmax following single dose of GSK2140944 | Up to Day 4
  Preliminary dose proportionality will be assessed using PK parameter Cmax following single dose of GSK2140944
Pharmacokinetic parameter: (Ae) following single dose of GSK2140944 | Up to Day 4
  Pharmacokinetic data will include urinary recovery of unchanged drug (Ae) following single dose of GSK2140944
Pharmacokinetic parameter: (CLr) following single dose of GSK2140944 | Up to Day 4
  Pharmacokinetic data will include renal clearance (CLr) following single dose of GSK2140944

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Tiffany C, Dumont EF, Hossain M, Srinivasan M, Swift B. Pharmacokinetics, safety, and tolerability of gepotidacin administered as single or repeat ascending doses, in healthy adults and elderly subjects. Clin Transl Sci. 2022 Sep;15(9):2251-2264. doi: 10.1111/cts.13359. Epub 2022 Jul 13. PMID 35769034
- See also: Results for study 114595 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/114595?search=study&search_terms=114595#rs